CLINICAL TRIAL: NCT06518408
Title: A Real-life Study of the Use of Cabotegravir Plus Rilpivirine Long-acting in ART-experienced Pre-treated People With HIV
Acronym: CABO-CHANCE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Virgen de las Nieves (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Carmen Hidalgo Tenorio, Professor, University Hospital Virgen de las Nieves
Other Study IDs: FIB-CAB-2023-02
Record Dates: First submitted 2024-07-09; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Long-Acting; Cabotegravir; Rilpivirine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — cabotegravir; Rilpivirine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- study group: Patients enrolled who switch to receive Cabotegravir long acting plus Rilpivirine long acting intramuscular injection every 2 months
  Interventions: Drug: Cabotegravir Injectable Product; Drug: Rilpivirine Injectable Product

INTERVENTIONS:
Drug: Cabotegravir Injectable Product — long-acting regimen dosed every 2-months
  Other Names: VOCABRIA (cabotegravir)
Drug: Rilpivirine Injectable Product — long-acting regimen dosed every 2-months
  Other Names: REKAMBYS (rilpivirine)

SUMMARY:
The CABOTEGRAVIR Long Acting + RILPIVIRENE Long Acting regimen was currently endorsed by guidelines worldwide as an option for the Treatment of HIV-1 Infection, however collecting real-world data closer to clinical practice use is still necessary. This study also registers some immunological, metabolic,anti-inflammatory parameters and fat distribution analysis to observe a hypothetical improvement on these parameters.

Psychosocial aspects are also very important in these patients as these patients may suffer social stigma, and therefore suffer certain psychological disorders. Patient experience data will be assessed through PROs and bespoke single-item questions to collect patient perception of treatment and register psychosocial aspects related to their health status.

ELIGIBILITY:
Inclusion Criteria: participants are required to meet all the following inclusion criteria to be eligible for PWH.

* Aged 18 years or older at the time of signing the informed consent.
* Virologically suppressed (HIV-1 RNA <50 copies/mL) on a stable antiretroviral regimen
* Documented evidence of plasma HIV-1 RNA measurements <50 copies/mL in the 6 months prior to Screening (1x blip is allowed).
* Ability to understand informed consent form (ICF) and other relevant regulatory documents.
* Prior to starting CAB LA + RPV LA injections, HIV physicians should have carefully selected patients who agree to the required injection schedule and counsel patients about the importance of adherence to scheduled dosing visits to help maintain viral suppression and reduce the risk of viral rebound and potential development of resistance with missed doses.
* A female subject is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine hCG test ) and not lactating. Females of childbearing potential will be required to use a highly effective method of contraception.

Exclusion Criteria: participants will be excluded from the trial if there is evidence of any of the following criteria at screening or check-in, as appropriate.

* Within 6 months prior to Screening, any plasma HIV-1 RNA measurement ≥50 copies/mL or within the 6 to 12-month window prior to Screening, any plasma HIV-1 RNA measurement >200 copies/mL, or 2 or more plasma HIV-1 RNA measurements ≥50 copies/mL.
* Previous antiretroviral treatment interruption during the last 6 months or treatment interruptions for more than a month.
* Present or past evidence of viral resistance to agents of the NNRTI or INI class or prior treatment failure with agents of NNRTI or INSTI class
* Any contraindication for CAB LA, RPV LA, oral Cabotegravir or Rilpivirine (see EU SmPC).
* Evidence of Hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (anti-HBc), Hepatitis B surface antibody (anti-HBs) and HBV DNA as follows:

  * Participants positive for HBsAg are excluded.
  * Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status), whether negative or positive for HBV DNA, are excluded.
  * Note: Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.
  * Participants treated with entecavir are not excluded.
* Any condition that does not recommend intramuscular injections in the gluteal muscle.
* Pregnancy or breastfeeding women, or with the desire to become pregnant soon.
* Current use of concomitant treatment with prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Virologically suppressed PWH, who switch to CAB LA + RPV LA Q2M (EU SmPC) from June 2023 to March 2024. Participants must meet all inclusion and no exclusion criteria. CAB LA + RPV LA injection may be preceded by an optional oral lead-in (OLI) according to the physician's judgement for 28 days
Sampling Method: Non-Probability Sample
Enrollment: 287 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants switching treatment to CAB LA + RPV LA regimen dosed every 2-months with plasma HIV-1 RNA ≥50 at month 12 | 12 months
  Proportion of participants suppressed on stable oral ART that switched to CAB LA + RPV LA with plasma HIV-1 RNA ≥50 copies/mL at month 12

SECONDARY OUTCOMES:
Number of participants switching treatment to CAB LA + RPV LA regimen dosed every 2-months with plasma HIV-1 RNA ≥50 at month 24 | 24 months
  Proportion of participants suppressed on stable oral ART that switch to CAB LA + RPV LA with plasma HIV-1 RNA ≥50 copies/mL at month 24
Number of participants switching treatment to CAB LA + RPV LA regimen dosed every 2-months with plasma HIV-1 RNA ≥50 at months 12 and 24 | 12 and 24 months
  Proportion of participants suppressed on stable oral ART that switch to CAB LA + RPV LA with plasma HIV-1 RNA <50 copies/mL at months 12 and 24
Number of episodes of plasma HIV-1 RNA ≥50 copies/mL | 24 months
  Number of episodes of plasma HIV-1 RNA ≥50 copies/mL that do not meet the criteria for confirmed virological failure
Number of participants experiencing confirmed virologic failure at months 12 and 24. | 12 and 24 months
  Proportion of participants experiencing confirmed virologic failure (CVF: two consecutive plasma HIV-1 RNA ≥200 copies/mL) at months 12 and 24.
Change from baseline in the mean lymphocyte subpopulations | 12 and 24 months
  Changes from baseline in the mean values of CD4, CD8 and CD4/CD8 ratio of participants switching to CAB LA + RPV LA at months 12 and 24.
Incidence and severity of adverse events | 24 months
  Proportion of emergence of adverse events, laboratory abnormalities and discontinuation rates due to adverse events. Includes severity evaluation of those
Description of reasons for discontinuation from CAB LA + RPV LA over 24 months | 24 months
  Reasons recorded for discontinuation of the study intervention during the follow-up
Number of reports fo adverse events over 24 months | 24 months
  Persistence over 24 months of adverse events, including injection site reactions (ISR), after switching to CAB LA + RPV LA
Description of reasons for switching to CAB LA + RPV LA | 24 months
  Reasons recorded for switching to the study intervention
Changes in absolute values from baseline over 24 months in metabolic control parameters: glucose | 24 months
  changes from baseline over 24 months and the proportion by patient subgroup with significant changes: in metabolic control parameters: glucose
Changes in absolute values from baseline over 24 months in metabolic control parameters: lipids | 24 months
  changes from baseline over 24 months and the proportion by patient subgroup with significant changes: in metabolic control parameters: lipids.
Changes in absolute values from baseline over 24 months in metabolic control parameters: weight | 24 months
  changes from baseline over 24 months and the proportion by patient subgroup with significant changes: in metabolic control parameters: weight.
Changes in absolute values from baseline over 24 months in metabolic control parameters: waist circumference. | 24 months
  changes from baseline over 24 months and the proportion by patient subgroup with significant changes: in metabolic control parameters: waist circumference.
Changes in absolute values from baseline over 24 months in metabolic control parameters: BMI | 24 months
  changes from baseline over 24 months and the proportion by patient subgroup with significant changes in metabolic control parameters: BMI (kg/m^2).
Changes in pro-inflammatory biomarkers (D-Dimmer) from baseline over 24 months in a subgroup of participants | 24 months
  Assesment and description in a subgroup of study participants of the change of pro-inflammatory biomarkers (D-Dimmer) after switching to CAB LA+ RPV LA through the study.
Changes in pro-inflammatory biomarkers (fibrinogen) from baseline over 24 months in a subgroup of participants | 24 months
  Assesment and description in a subgroup of study participants of the change of pro-inflammatory biomarkers (fibrinogen) after switching to CAB LA+ RPV LA through the study.
Changes in pro-inflammatory biomarkers (CRP) from baseline over 24 months in a subgroup of participants | 24 months
  Assesment and description in a subgroup of study participants of the change of pro-inflammatory biomarkers (CRP) after switching to CAB LA+ RPV LA through the study.
Changes in pro-inflammatory biomarkers (IL-6) from baseline over 24 months in a subgroup of participants | 24 months
  Assesment and description in a subgroup of study participants of the change of pro-inflammatory biomarkers (IL-6) after switching to CAB LA+ RPV LA through the study.
Changes in creatinine values from baseline over 24 months | 24 months
  Changes from baseline over 24 months in creatinine (mg/dL) values after switching to CAB LA + RPV LA
Changes in hepatic values (Albumine) from baseline over 24 months | 24 months
  Changes from baseline over 24 months in hepatic values (Albumine) in g/dL after switching to CAB LA + RPV LA
Changes in hepatic values (Alanine transaminase (ALT), Aspartate transaminase (AST) and Alkaline phosphatase (ALP)) from baseline over 24 months | 24 months
  Changes from baseline over 24 months in hepatic values (Alanine transaminase (ALT), Aspartate transaminase (AST) and Alkaline phosphatase (ALP)) in U/L after switching to CAB LA + RPV LA
Changes in preference values from baseline over 24 months about ART | 12 and 24 months
  Rate of ART preference of LA-injected vs. oral ART at months12 and 24 and description of reasons
Changes in patient reported outcomes questionnaires from baseline over 24 months: WHOQOL-HIV-BREF | 24 months
  Changes from baseline in domains of PROs: World Health Organization Quality of Life, on Human Immunodeficiency Virus, brief version (WHOQOL-HIV-BREF) scale over 24 months and the proportion by patient subgroup with significant changes. MIN VALUE 26- MAX VALUE 130. Higher scores mean better quality of life.
Changes in patient reported outcomes questionnaires from baseline over 24 months: HSSS | 24 months
  Changes from baseline in domains of PROs: adapted HIV Stigma Scale for use in Spain (HSSS) scale over 24 months and the proportion by patient subgroup with significant changes. Scores can range from 40 to 160 [1 x 40 items to 4 x 40 items]. Higher scores indicate greater feelings of stigma
Changes in patient reported outcomes questionnaires from baseline over 24 months: PSQI | 24 months
  Changes from baseline in domains of PROs: Pittsburgh Sleep Quality Index (PSQI) scale over 24 months and the proportion by patient subgroup with significant changes. Score has a possible range of 0-21 points. Higher scores means better sleep quality
Incidence of adherence to scheduled interventions over 24 months | 24 months
  * Number and percentage of total injections within ±7-day dosing window
  * Number and percentage of missed injections.

CONTACTS AND LOCATIONS:
Overall Officials: CARMEN HIDALGO, PhD, Principal Investigator — HU Virgen de las Nieves
Locations (15):
- Spain (15):
  - Hospital Universitario Virgen de Las Nieves, Granada, Andalusia
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Reina Sofía, Murcia, Murcia
  - Hospital Universitario Puerto Real, INIBICA,, Cadiz
  - Jerez de la Frontera University Hospital, Cadiz
  - Reina Sofía University Hospital, Córdoba
  - Hospital Campus de la Salud, Granada
  - Hospital Comarcal Santa Ana de Motril, Granada
  - Complejo Hospitalario de Jaén,, Jaén
  - Hu La Princesa, Madrid
  - Ramon Y Cajal, Madrid
  - Hospital General Universitario Santa Lucía, Murcia
  - Hospital de Son Llàtzer, Palma de Mallorca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza